CLINICAL TRIAL: NCT03959527
Title: A Multi-center, Randomized, Open-label, Non Inferiority Trial to Evaluate the Efficacy and Safety of a Single, Oral Dose of Zoliflodacin Compared to a Combination of a Single Intramuscular Dose of Ceftriaxone and a Single Oral Dose of Azithromycin in the Treatment of Patients With Uncomplicated Gonorrhoea
Brief Title: Zoliflodacin in Uncomplicated Gonorrhoea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Global Antibiotics Research and Development Partnership (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STI_Zoli001; 2019-000990-22 (EudraCT Number)
Record Dates: First submitted 2019-05-02; First posted 2019-05-22 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Gonorrhea
MeSH Terms: conditions — Gonorrhea | interventions — zoliflodacin; Ceftriaxone; Azithromycin

STUDY DESIGN:
Intervention Model Description: Single dose of Zoliflodacin or comparators combination in single dose: ceftriaxone and azithromycin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- zoliflodacin (Experimental): Participant in this arm will receive a single dose of zoliflodacin.
  Interventions: Drug: zoliflodacin
- ceftriaxone and azithromycin combination (Active Comparator): Participant in this arm will receive a single dose of comparators combination (ceftriaxone and azithromycin).
  Interventions: Drug: ceftriaxone; Drug: azithromycin

INTERVENTIONS:
Drug: zoliflodacin — Dose: 3g, oral administration
  Arms: zoliflodacin
Drug: ceftriaxone — Dose: 500mg, Intra-Muscular (IM) administration
  Arms: ceftriaxone and azithromycin combination
Drug: azithromycin — Dose: 1g, oral administration
  Arms: ceftriaxone and azithromycin combination

SUMMARY:
This trial is a multi-center, open label, randomized controlled, non-inferiority phase III trial evaluating the safety and efficacy of a 3 g oral dose of zoliflodacin compared to a combination of a single intra-muscular 500 mg dose of ceftriaxone and a single 1 g oral dose of azithromycin for the treatment of uncomplicated gonorrhoea.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12 years old (if enrolment of minors is in agreement with local regulations and Ethics guidance)
2. Weight ≥ 35 kg
3. Signs and symptoms consistent with urethral or cervical gonorrhoea OR Urethral or cervical uncomplicated gonorrhoea as determined by either a positive culture or NAAT or Gram stain or methylene blue test/gentian violet stain in the past 14 days prior to screening OR Unprotected sexual contact with an individual reported to be infected with NG in the past 14 days prior to screening (confirmation by a positive NAAT, Gram stain or methylene blue test/ gentian violet stain or culture)
4. For females of child-bearing potential, a negative urine pregnancy test at screening
5. For females of child bearing potential, use of highly effective contraception for at least 28 days prior to screening and during at least 28 days after treatment. Females on oral contraceptives must also use a barrier contraception method during participation in the study.
6. For males with a female partner of child-bearing age, willingness to delay conception for 28 days after treatment
7. Willingness to comply with trial protocol
8. Willingness to undergo HIV testing
9. Willingness to abstain from sexual intercourse or use condoms for vaginal, anal and oral sex until end of trial visit
10. Willingness and ability to give written informed consent or be consented by a legal representative or provide assent and parental consent (for minors, as appropriate).

    Exclusion Criteria:
11. Confirmed or suspected complicated or disseminated gonorrhoea
12. Pregnant or breastfeeding women
13. Known concomitant infection which would require immediate additional systemic antibiotics with activity against NG (e.g. CT infection)
14. Use of any systemic or intravaginal antibiotics with activity against NG within 30 days prior to screening
15. Use of systemic corticoid drugs or other immunosuppressive therapy within 30 days prior to screening
16. Use of moderate or strong CYP3A4 inducers (e.g. efavirenz, rifampicin, carbamazepine, phenobarbital) within 30 days or five half-lives of the drug, whichever is greater, prior to screening
17. Cytotoxic or radiation therapy within 30 days prior to screening
18. Known chronic renal, hepatic, hematologic impairment or other condition interfering with the absorption, distribution or elimination of the drug based on medical history and physical examination
19. History of urogenital sex-reassignment surgery
20. Immunosuppression as evidenced by medical history, clinical examination or a recent (≤ 1 month) CD4 count <200 cells/μL
21. Know clinically relevant cardiac pro-arrhythmic conditions such as cardiac arrhythmia, congenital or documented QT prolongation
22. Known history of severe allergy to cephalosporin, penicillin, monobactams, carbapenems or macrolide antibiotics
23. Known or suspected allergies or hypersensitivities to lidocaine, methylparaben, lactose or any of the components of the study drugs (refer to the zoliflodacin IB and SmPC for the comparators treatments)
24. Receipt or planned receipt of an investigational product in a clinical trial within 30 days or five half-lives of the drug, whichever is greater, prior to screening until end of participation to this clinical trial
25. History of alcohol or drug abuse within 12 months prior to screening which would compromise trial participation in the judgment of the investigator
26. Severe medical or psychiatric condition which, in the opinion of the investigator, may increase the risk associated with trial participation or may interfere with the interpretation of trial results or affect the individual's ability to provide informed consent
27. Individuals whom, in the judgement of the investigator, are unlikely or unable to comply with this trial protocol
28. Previous randomisation in this clinical trial.
29. Use of moderate or strong CYP3A4 inhibitors within 30 days or five half-lives of the drug, whichever is greater, prior to screening

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1011 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (6):
  - Jefferson County Department of Health, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - San Francisco Department Of Public Health City Clinic, San Francisco, California
  - Bell Flower Clinic, Indianapolis, Indiana
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Public Health - Seattle & King County STD Clinic, Seattle, Washington
- Institute of Tropical Medicine, Antwerp, Belgium
- Public Health Service (GGD) Amsterdam / STI Outpatient Clinic, Amsterdam, Netherlands
- South Africa (6):
  - SAMRC Botha's Hill Clinical Research Site, Bothas Hill
  - Masiphumelele Research Site, Cape Town
  - Ndlovu Research Centre, Elandsdoorn
  - Wits RHI, Johannesburg
  - Setshaba Research Centre, Soshanguve
  - SAMRC Tongaat Clinical Research Site, Tongaat
- Thailand (3):
  - Bangrak STI Center, Bangkok
  - Institute of HIV Research and Innovation, Bangkok
  - Silom Community Clinic, Bangkok

REFERENCES:
- [Derived] Luckey A, Balasegaram M, Barbee LA, Batteiger TA, Broadhurst H, Cohen SE, Delany-Moretlwe S, de Vries HJC, Dionne JA, Gill K, Kenyon C, Kittiyaowamarn R, Lewis D, Mueller JP, Naicker V, O'Brien S, O'Donnell JP, Phanuphak N, Spooner E, Srinivasan S, Taylor SN, Unemo M, Zwane Z, Hook EW 3rd; Zoliflodacin Phase 3 Study Group. Zoliflodacin versus ceftriaxone plus azithromycin for treatment of uncomplicated urogenital gonorrhoea: an international, randomised, controlled, open-label, phase 3, non-inferiority clinical trial. Lancet. 2026 Jan 10;407(10524):147-160. doi: 10.1016/S0140-6736(25)01953-1. Epub 2025 Dec 11. PMID 41391465
- [Derived] Jacobsson S, Golparian D, Oxelbark J, Kong FYS, Da Costa RMA, Franceschi F, Brown D, Louie A, Drusano G, Unemo M. Pharmacodynamics of zoliflodacin plus doxycycline combination therapy against Neisseria gonorrhoeae in a gonococcal hollow-fiber infection model. Front Pharmacol. 2023 Dec 7;14:1291885. doi: 10.3389/fphar.2023.1291885. eCollection 2023. PMID 38130409

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 1011 participants were screened, of which 81 were screen failure
Period: Overall Study
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination
Started | 621 | 309
Completed | 571 | 285
Not Completed | 50 | 24
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Lost to Follow-up | 31 | 15
Not completed — Did not meet eligibility criteria | 1 | 1
Not completed — Protocol Violation | 10 | 5

BASELINE CHARACTERISTICS:
Population: Randomised population
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination | Total
Number analyzed (Participants) | 621 | 309 | 930
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (9.56) | 29.2 (9.13) | 29.7 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 38 | 115
  Male | 544 | 271 | 815
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 13 | 31
  Not Hispanic or Latino | 603 | 296 | 899
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 1 | 9
  Asian | 193 | 92 | 285
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 349 | 165 | 514
  White | 66 | 47 | 113
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Netherlands | 49 | 20 | 69
  Belgium | 6 | 3 | 9
  United States | 107 | 51 | 158
  South Africa | 278 | 146 | 424
  Thailand | 181 | 89 | 270

OUTCOME MEASURES:

1. Primary Outcome: Microbiological Cure Rate for Zoliflodacin Compared to a Combination of a Single Dose of Ceftriaxone and Azithromycin.
Description: Proportion of participants with microbiological cure as determined by culture at urethral or cervical sites at test of cure visit in micro-ITT (urogenital) analysis set
Time Frame: Day 6 (+/- 2)
Population: micro-ITT (urogenital): all randomized participants who had a positive NG culture from the relevant anatomical site at baseline and whose baseline AST result showed no pre-existing resistance to both ceftriaxone and azithromycin
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination
Number analyzed (Participants) | 506 | 238
percentage of participants | 90.9 [88.1 to 93.3] | 96.2 [92.9 to 98.3]
Statistical Analysis 1: Comparison: Zoliflodacin vs Ceftriaxone and Azithromycin Combination; Point estimate for the treatment difference in proportion of ceftriaxone/azithromycin combination and zoliflodacin with microbiological cure and 2-sided 95% CI calculated by Newcombe score method; Test type: Non-Inferiority — A single oral 3 g dose of zoliflodacin would be considered as non-inferior to a combination of a single IM 500 mg dose of ceftriaxone and a single 1 g oral dose of azithromycin if the upper bound of the 2-sided 95% CI for the microbiological cure rate of the combination therapy minus zoliflodacin was less than 12% (prespecified non-inferiority [NI] margin for the primary endpoint); Risk Difference (RD) = 5.31, 95% CI 2-sided [1.38 to 8.65] — 95% CI of the treatment difference of ceftriaxone+ azithromycin combination minus zoliflodacin

2. Secondary Outcome: Safety of a Single Dose of Zoliflodacin Will be Assessed Compared to a Combination a Single Dose of Ceftriaxone and Azithromycin.
Description: Incidence, severity, causality and seriousness of treatment-emergent adverse events (including clinically significant abnormal laboratory values/procedures i.e., physical examination per protocol)
Time Frame: Day 30
Population: The safety population included all randomized participants who received any part of trial treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination
Number analyzed (Participants) | 619 | 308
Participants
  All AEs | 287 | 144
  Related AEs | 117 | 76
  Serious AEs | 0 | 0
  AEs leading to treatment discontinuation | 0 | 0
  AEs leading to death | 0 | 0
  Maximum severity CTCAE Grade 1 or Mild | 157 | 82
  Maximum severity CTCAE Grade 2 or Moderate | 109 | 44
  Maximum severity CTCAE Grade 3 or Severe | 20 | 18
  Maximum severity CTCAE Grade 4 or Life-Threatening | 1 | 0
  Maximum severity CTCAE Grade 5 or Death | 0 | 0

3. Secondary Outcome: Microbiological Cure Rate of Pharyngeal Gonorrhoea of a Single Dose of Zoliflodacin Compared to a Single Dose of Ceftriaxone and Azithromycin.
Description: Proportion of participants with microbiological cure as determined by NG culture at pharyngeal sites at test of cure visit in micro-ITT (Pharyngeal).
Time Frame: Day 6
Population: Micro-ITT (Pharyngeal) population: all randomized participants who had a positive NG culture from the pharyngeal site at baseline and whose baseline AST result showed no pre-existing resistance to both ceftriaxone and azithromycin
Measure: Count of Participants; unit: Participants
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination
Number analyzed (Participants) | 53 | 28
Participants | 42 | 22

4. Secondary Outcome: Microbiological Cure Rate of Rectal Gonorrhoea of a Single Dose of Zoliflodacin Compared to a Single Dose of Ceftriaxone and Azithromycin.
Description: Proportion of participants with microbiological cure as determined by NG culture at rectal sites at test of cure visit in micro-ITT (Rectal).
Time Frame: Day 6
Population: Micro-ITT (Rectal): all randomized participants who had a positive NG culture from the rectal site at baseline and whose baseline AST result showed no pre-existing resistance to both ceftriaxone and azithromycin
Measure: Count of Participants; unit: Participants
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination
Number analyzed (Participants) | 79 | 35
Participants | 69 | 31

5. Secondary Outcome: The Clinical Cure Rate in Male Participants After Administration of a Single Dose of Zoliflodacin Compared to a Single Dose of Ceftriaxone and Azithromycin.
Description: Proportion of male at birth participants experiencing resolution of signs and symptoms of urogenital gonococcal infection that were present at enrolment, at test of cure visit in Clinical Cure Population.
Time Frame: Day 6
Population: Clinical Cure population: all participants assigned male at birth included in the Micro-ITT (urogenital) population and who had at least one sign or symptom of urethral gonorrhea at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination
Number analyzed (Participants) | 460 | 220
Participants | 375 | 194

6. Secondary Outcome: Microbiological Cure Rate Among Females, After Administration of a Single Dose of Zoliflodacin Compared to a Single Dose of Ceftriaxone and Azithromycin
Description: Proportion of female participants with microbiological cure, as determined by NG culture at cervical site of infection, at TOC in micro-ITT (Urogenital) population
Time Frame: Day 6
Population: micro-ITT (Urogenital): all randomized participants who had a positive NG culture from the urogenital site at baseline and whose baseline AST result showed no pre-existing resistance to both ceftriaxone and azithromycin
Measure: Count of Participants; unit: Participants
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination
Number analyzed (Participants) | 50 | 18
Participants | 48 | 16

7. Secondary Outcome: Microbiological Cure Rate Among Males, After Administration of a Single Dose of Zoliflodacin Compared to a Single Dose of Ceftriaxone and Azithromycin
Description: Proportion of male participants with microbiological cure as determined by NG culture at urethral site of infection at TOC visit, in micro-ITT population
Time Frame: Day 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination
Number analyzed (Participants) | 456 | 220
Participants | 412 | 213

8. Secondary Outcome: Eradication of Urogenital NG NAAT at TOC After Administration of a Single Dose of Zoliflodacin Compared to a Single Dose of Ceftriaxone and Azithromycin.
Description: Proportion of participants with a positive NG NAAT result from urethral or cervical sites at baseline and a negative NG NAAT result at test of cure visit in micro-ITT analysis set.
Time Frame: Day 6
Population: Of those participants included in the micro-ITT (Urogenital) analysis set (i.e., all randomized participants who had a positive NG culture from the urogenital site at baseline and whose baseline AST result showed no pre-existing resistance to both ceftriaxone and azithromycin) (N=744), a total of 725 had a positive NG NAAT result at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination
Number analyzed (Participants) | 492 | 233
Participants | 405 | 190

9. Secondary Outcome: Eradication of Pharyngeal NG NAAT at TOC After Administration of a Single Dose of Zoliflodacin Compared to a Single Dose of Ceftriaxone and Azithromycin.
Description: Proportion of participants with a positive NG NAAT at baseline from pharyngeal sites and a negative NG NAAT at test of cure visit in micro-ITT analysis set.
Time Frame: Day 6
Population: Of those participants included in the micro-ITT (Pharyngeal) analysis set (N=81) (i.e., all randomized participants who had a positive NG culture from the pharyngeal site at baseline and whose baseline AST result showed no pre-existing resistance to both ceftriaxone and azithromycin), a total of 69 had positive pharyngeal NG NAAT result
Measure: Count of Participants; unit: Participants
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination
Number analyzed (Participants) | 45 | 24
Participants | 28 | 12

10. Secondary Outcome: Eradication of Rectal NG NAAT at TOC After Administration of a Single Dose of Zoliflodacin Compared to a Single Dose of Ceftriaxone and Azithromycin.
Description: Proportion of participants with a positive NG NAAT from rectal sites at baseline and a negative NG NAAT at test of cure visit in micro-ITT analysis set.
Time Frame: Day 6
Population: Of those participants included in the micro-ITT (Rectal) analysis set (N=114) (i.e., all randomized participants who had a positive NG culture from the rectal site at baseline and whose baseline AST result showed no pre-existing resistance to both ceftriaxone and azithromycin), a total of 103 had a positive NG NAAT result at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination
Number analyzed (Participants) | 73 | 30
Participants | 60 | 27

11. Secondary Outcome: Arithmetic Mean Plasma Concentration of Zoliflodacin
Description: Arithmetic mean plasma concentration (ng/mL) of zoliflodacin following oral administration of single oral dose of zoliflodacin 3 g
Time Frame: 15 min - 1 hour
Population: Of the 23 participants included in the PK Population Set (all participants randomized to the zoliflodacin group who consent to participate to the PK sub-trial and from whom at least one valid PK sample post treatment is obtained), quantifiable zoliflodacin concentrations were available for only 22 participants at this time point
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 22
ng/mL | 580 (830)

12. Secondary Outcome: Arithmetic Mean Plasma Concentration of Zoliflodacin
Description: Arithmetic mean plasma concentration (ng/mL) of zoliflodacin following a single oral dose administration of zoliflodacin 3 g
Time Frame: 2-2.5 h
Population: PK Population Set (all participants randomized to the zoliflodacin group who consent to participate to the PK sub-trial and from whom at least one valid PK sample post treatment is obtained).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 23
ng/mL | 14500 (9610)

13. Secondary Outcome: Arithmetic Mean Plasma Concentration of Zoliflodacin
Description: Arithmetic mean plasma concentration (ng/mL) of zoliflodacin following administration of a single oral dose of zoliflodacin 3 g
Time Frame: 4.5 - 5h
Population: The PK population will include all participants randomized to the zoliflodacin group who consent to participate to the PK sub-trial and from whom at least one valid PK sample post treatment is obtained.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 23
ng/mL | 32300 (8630)

14. Secondary Outcome: Arithmetic Mean Plasma Concentration of Zoliflodacin
Description: Arithmetic mean plasma concentration (ng/mL) of zoliflodacin following administration of a single oral dose zoliflodacin 3 g
Time Frame: 10 -12 h
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 23
ng/mL | 19300 (6000)

15. Secondary Outcome: Arithmetic Mean Plasma Concentration of Zoliflodacin
Description: as for outcome 13
Time Frame: 24 - 36 h
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 23
ng/mL | 3270 (1560)

16. Secondary Outcome: Evaluation of the Plasma PK Profile (Tlast) After a Single, Oral, 3 g Dose of Zoliflodacin
Description: Geometric mean time to last (Tlast) plasma concentration above the lower limit of quantitation
Time Frame: Day 2
Population: PK population: all participants randomized to the zoliflodacin group who consent to participate to the PK sub-trial and from whom at least one valid PK sample post treatment is obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 23
hours | 24.6 (3.2)

17. Secondary Outcome: Evaluation of the Plasma PK Profile(Tmax) After a Single, Oral, 3 g Dose of Zoliflodacin
Description: Geometric mean time to maximum plasma concentration (Tmax) after a single, oral, 3 g dose of zoliflodacin
Time Frame: Day 2
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 23
hours | 4.83 (41.0)

18. Secondary Outcome: Evaluation of the Plasma PK Profile (Cmax) After a Single, Oral, 3 g Dose of Zoliflodacin
Description: Geometric mean maximum plasma concentration (Cmax) after a single, oral 3 g dose of zoliflodacin
Time Frame: Day 2
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 23
ng/mL | 31800 (27.3)

19. Secondary Outcome: Evaluation of the Plasma PK Profile After a Single, Oral, 3 g Dose of Zoliflodacin
Description: Geometric mean plasma area under the concentration-time curve (AUC0-last) from time zero to the last concentration above lower level of quantification
Time Frame: Day 2
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 23
h*ng/mL | 330000 (26.5)

20. Secondary Outcome: Antimicrobial Susceptibility (Azithromycin) Profile of NG Isolates Obtained at Baseline (Day 1)
Description: Antimicrobial susceptibility to azithromycin (MIC90) - profile of gonococcal strains isolated from urogenital site at baseline (Day 1)
Time Frame: Day 1
Population: Number of participants in urogenital micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Groups:
- Ceftriaxone Plus Azithromycin Combination: Participant in this arm will receive a single dose of comparators combination (ceftriaxone and azithromycin).
  ceftriaxone: Dose: 500mg, Intra-Muscular (IM) administration
  azithromycin: Dose: 1g, oral administration
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 506 | 238
mg/L | 1 [0.06 to 8] | 1 [0.06 to 8]

21. Secondary Outcome: Antimicrobial Susceptibility (Azithromycin) Profile of NG Isolates Obtained at Test of Cure Visit.
Description: Antimicrobial susceptibility to azithromycin (MIC90) - profile of gonococcal strains isolated from urogenital site at TOC
Time Frame: Day 6
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 15 | 0
mg/L | 0.25 [0.06 to 2] |

22. Secondary Outcome: Antimicrobial Susceptibility (Cefixime) Profile of NG Isolates Obtained at Baseline
Description: Antimicrobial susceptibility to cefixime (MIC90) - profile of gonococcal strains isolated from urogenital site at baseline
Time Frame: Day 1
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 506 | 238
mg/L | 0.06 [0.002 to 0.5] | 0.06 [0.002 to 0.5]

23. Secondary Outcome: Antimicrobial Susceptibility (Cefixime) Profile of NG Isolates Obtained at Test of Cure Visit.
Description: Antimicrobial susceptibility to cefixime (MIC90) - profile of gonococcal strains isolated from urogenital site at TOC
Time Frame: Day 6
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 15 | 0
mg/L | 0.015 [0.002 to 0.03] |

24. Secondary Outcome: Antimicrobial Susceptibility (Ceftriaxone) Profile of NG Isolates Obtained at Baseline
Description: Antimicrobial susceptibility to ceftriaxone (MIC90) - profile of gonococcal strains isolated from urogenital site at baseline
Time Frame: Day 1
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 506 | 238
mg/L | 0.015 [0.002 to 0.25] | 0.015 [0.002 to 0.12]

25. Secondary Outcome: Antimicrobial Susceptibility (Ceftriaxone) Profile of NG Isolates Obtained at Test of Cure Visit.
Description: Antimicrobial susceptibility to ceftriaxone (MIC90) - profile of gonococcal strains isolated from urogenital site at TOC
Time Frame: Day 6
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 15 | 0
mg/L | 0.015 [0.002 to 0.015] |

26. Secondary Outcome: Antimicrobial Susceptibility (Ciprofloxacin) Profile of NG Isolates Obtained at Baseline
Description: Antimicrobial susceptibility to ciprofloxacin (MIC90) - profile of gonococcal strains isolated from urogenital site at baseline (zoliflodacin arm only since no microbiological failures in comparator arm)
Time Frame: Day 1
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 506 | 238
mg/L | 2 [0.0005 to 2] | 2 [0.002 to 2]

27. Secondary Outcome: Antimicrobial Susceptibility (Ciprofloxacin) Profile of NG Isolates Obtained at Test of Cure Visit
Description: as for outcome 21
Time Frame: Day 6
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 15 | 0
mg/L | 2 [0.004 to 2] |

28. Secondary Outcome: Antimicrobial Susceptibility (Gentamicin) Profile of NG Isolates Obtained at Baseline
Description: Antimicrobial susceptibility to gentamicin (MIC90) - profile of gonococcal strains isolated from urogenital site at baseline
Time Frame: Day 1
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 506 | 238
mg/L | 8 [1 to 16] | 8 [0.5 to 16]

29. Secondary Outcome: Antimicrobial Susceptibility (Gentamicin) Profile of NG Isolates Obtained at Test of Cure Visit.
Description: Antimicrobial susceptibility to gentamicin (MIC90) - profile of gonococcal strains isolated from urogenital site at TOC
Time Frame: Day 6
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 15 | 0
mg/L | 8 [4 to 8] |

30. Secondary Outcome: Antimicrobial Susceptibility (Spectinomycin) Profile of NG Isolates Obtained at Baseline
Description: Antimicrobial susceptibility to spectinomycin (MIC90) - profile of gonococcal strains isolated from urogenital site at baseline
Time Frame: Day 1
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 506 | 238
mg/L | 32 [8 to 64] | 32 [8 to 64]

31. Secondary Outcome: Antimicrobial Susceptibility (Spectinomycin) Profile of NG Isolates Obtained at Test of Cure Visit
Description: Antimicrobial susceptibility to spectinomycin (MIC90) - profile of gonococcal strains isolated from urogenital site at TOC
Time Frame: Day 6
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 15 | 0
mg/L | 32 [16 to 32] |

32. Secondary Outcome: Antimicrobial Susceptibility (Tetracycline) Profile of NG Isolates Obtained at Baseline
Description: Antimicrobial susceptibility to tetracycline (MIC90) - profile of gonococcal strains isolated from urogenital site at baseline
Time Frame: Day 1
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 506 | 238
mg/L | 4 [0.12 to 4] | 4 [0.12 to 4]

33. Secondary Outcome: Antimicrobial Susceptibility (Tetracycline) Profile of NG Isolates Obtained at Test of Cure Visit
Description: Antimicrobial susceptibility to tetracycline (MIC90) - profile of gonococcal strains isolated from urogenital site at TOC
Time Frame: Day 6
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 15 | 0
mg/L | 4 [0.5 to 4] |

34. Secondary Outcome: Antimicrobial Susceptibility (Zoliflodacin) Profile of NG Isolates Obtained at Baseline
Description: Antimicrobial susceptibility to zolflodacin (MIC90) - profile of gonococcal strains isolated from urogenital site at baseline
Time Frame: Day 1
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 506 | 238
mg/L | 0.12 [0.008 to 0.5] | 0.12 [0.008 to 0.25]

35. Secondary Outcome: Antimicrobial Susceptibility (Zoliflodacin) Profile of NG Isolates Obtained at Test of Cure Visit
Description: Antimicrobial susceptibility to zoliflodacin (MIC90) - profile of gonococcal strains isolated from urogenital site at TOC
Time Frame: Day 6
Population: Number of participants in urogenital Micro-ITT without missing data for the specified visit
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Zoliflodacin | Ceftriaxone Plus Azithromycin Combination
Number analyzed (Participants) | 15 | 0
mg/L | 0.12 [0.008 to 0.25] |

ADVERSE EVENTS:
Time Frame: 30 days (+/- 3 days)
Description: All adverse events (AE) that occurred between Day -1 to Day 30 are reported, irrespective of causality assessment. Any AE that occurs after the reporting period assessed as possibly related to the investigational treatment should also be reported.
  For screening failure participants, AEs are reported up until the date the participant was determined to be a screening failure. Beyond that date, only serious or medically relevant protocol-related events will be followed-up.
Arm/Group | Zoliflodacin | Ceftriaxone and Azithromycin Combination
All-Cause Mortality (participants affected / at risk) | 0/619 | 0/308
Serious Adverse Events (participants affected / at risk) | 0/619 | 0/308
Other Adverse Events (participants affected / at risk) | 162/619 | 107/308
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoliflodacin (N=619) | Ceftriaxone and Azithromycin Combination (N=308)
Neutropenia (Blood and lymphatic system disorders) | 42 (42) | 24 (24)
Leukopenia (Blood and lymphatic system disorders) | 24 (24) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 15 (15) | 22 (22)
Nausea (Gastrointestinal disorders) | 16 (16) | 12 (13)
Injection site pain (General disorders) | 5 (6) | 38 (38)
Neutrophil count decreased (Investigations) | 21 (21) | 15 (15)
Headache (Nervous system disorders) | 61 (65) | 14 (15)
Dizziness (Nervous system disorders) | 21 (21) | 5 (5)

LIMITATIONS AND CAVEATS:
Relatively low representation of females in primary analysis set due to asymptomatic nature of NG in this population, non-specific symptoms and inclusion criteria (prior contraceptive use).

Relatively low representation of adolescents in study and non in PK sub-study, due to challenges with obtaining parental consent primarily in this indication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and can extend the embargo for a further 90 days in order to enable the sponsor to take steps to protect its proprietary information and/or Intellectual Property Rights.

DOCUMENTS (3):
  • Study Protocol (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT03959527/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT03959527/SAP_001.pdf
  • Informed Consent Form (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT03959527/ICF_003.pdf